CLINICAL TRIAL: NCT02271581
Title: INSYNC: Leo Jenkins Cancer Center (LJCC) - Symptom Management Service (SMS) Protocol -Phase II Trial Regarding The Effect Of Comprehensive Symptom Management On Inflammation And Survival In Metastatic Lung Cancer
Brief Title: Effect of Symptom Management on Inflammation and Survival in Metastatic Lung Cancer
Status: Completed | Type: Observational
Sponsor: Leo W. Jenkins Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: INSYNC
Record Dates: First submitted 2014-07-30; First posted 2014-10-22 (Estimated); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Lung Neoplasms; Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Retain serum samples draw at baseline, 4 months, 10 months for storage and analysis by Biodesix Laboratories.
Oversight: Data Monitoring Committee: No

SUMMARY:
There is a growing body of evidence that implicates inflammation as a mechanism of disease progression and reduced survival in patients with advanced cancer. Elevated c-reactive protein levels have been shown to be associated with reduced performance status, specific cancer related symptoms and reduced overall survival. C-reactive protein levels are a surrogate for IL-6 expression. IL-6 is part of an inflammatory signature predicting cancer recurrence. VeriStrat® is a multivariate test which measures protein expression related to a host/tumor interaction mediated by inflammation. The investigators hope to examine the relationship between quality of life outcomes per FACT-L survey and correlate them with changes in c-reactive protein levels and the VeriStrat® status. The hypothesis of this study is that the remarkable survival benefit in the Temel study is mediated by reduced inflammation with improvement of symptom control.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of stage IV non-small cell lung cancer
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Able to read and respond to questions in English

Exclusion Criteria:

* Small Cell Lung Cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with metastatic (stage IV) non-small cell lung cancer
Sampling Method: Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2014-10; Primary Completion 2019-04-19 (Actual); Study Completion 2019-04-19 (Actual)

PRIMARY OUTCOMES:
Overall Survival | Patients will be followed for 5 years after enrolling last patient
  Overall survival from diagnosis until death from any cause

SECONDARY OUTCOMES:
Percentage of patients who convert from c-reactive protein 'high' (> 10 mg/L) to 'low' (<10 mg/L) | 10 months
  1. Baseline versus 4 months
  2. Baseline versus 10 months
  3. 4 months versus 10 months
Quality of Life (QOL) indicators per FACT-L score and the following at baseline, 4 months and 10 months groups | 10 months
  1. VeriStrat "Good" and CRP "low" (<10 mg/L)
  2. VeriStrat "Good" and CRP "high" (>10 mg/L)
  3. VeriStrat "Poor" and CRP "low" (<10 mg/L)
  4. VeriStrat "Poor" and CRP "high" (>10 mg/L)
Change in VeriStrat status | 10 months
  Percentage of patients who convert from "poor" to "good"

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Stroud, PharmD, BCOP, CPP, Principal Investigator — Brody School of Medicine at ECU
Locations (1):
- Leo Jenkins Cancer Center, Greenville, North Carolina, United States